CLINICAL TRIAL: NCT06108128
Title: Characterizing Top-down Dimensions of Appetite Self-regulation Among Preschoolers
Brief Title: Food for Thought: Executive Functioning Around Eating Among Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Baylor College of Medicine (Other); University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Jennifer Orlet Fisher, Professor, Temple University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R21HD109362 (NIH)
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Self-regulation; Appetitive Behavior; Eating Behavior; Child Obesity
MeSH Terms: conditions — Self-Control; Appetitive Behavior; Feeding Behavior; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This is an observational, cross-sectional study that involves interventions ONLY at the measurement level.
Masking Description: This is an observational cross-sectional study with interventions ONLY at the measurement level. The research assistant administers the tasks and records the outcomes; therefore, no masking is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Executive functioning observational tasks — Interventions take place solely at the measurement level, where children will be seen in observational tasks of general executive functioning and executive functioning around eating in which various food and non-food stimuli are presented and children's responses to task instructions are recorded.

SUMMARY:
Scientific knowledge of the cognitive-developmental processes that serve to support children's appetite self-regulation are surprisingly limited. This investigation will provide new scientific directions for obesity prevention by elucidating cognitive-developmental influences on young children's ability to make healthy food choices and eat in moderation.

DETAILED DESCRIPTION:
Appetite self-regulation (ASR) has been described as involving children's use of eating-specific, "top-down" cognitive processes to moderate "bottom-up" biological drives to eat. Much of the research to date on ASR has focused on the role of bottom-up drives in shaping children's behavioral susceptibility to obesity. Alternatively, little is known about the cognitive-developmental processes that shape children's ability to make healthy food choices and eat in moderation during early childhood. The goal of this exploratory investigation is to produce rigorous evidence of cognitive developmental influences on healthy eating behaviors and weight status during preschool through the development of new measures of top-down ASR. Participants will be 125 preschoolers and their primary caregiver. Existing measures of executive functioning in children will be adapted to create new measures of eating-specific, top-down ASR. Associations with children's eating behaviors, body mass index z-scores, food parenting will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Child ages 4 to 6 years of age
2. Caregiver reporting primary responsibility for child feeding outside of childcare
3. Caregiver legal guardian

Exclusion Criteria:

1. Caregiver <18 years of age
2. Child major food allergies
3. Child medication use, developmental disability, or medical conditions known to affect food intake and/or growth; color blindness
4. Child in foster care

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Food choice | Assessed at 1 of 2 study visits over 2 weeks
  Children's forced-choice selection of fruits, vegetables, and water over alternatives at a meal
Eating in the absence of hunger | Assessed at 1 of 2 study visits over 2 weeks
  Children's intake of palatable foods following a standard meal
Body mass index z-score | Assessed at 1 of 2 study visits over 2 weeks
  Age and sex specific z-score using CDC reference data

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer O Fisher, PHD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data generated by the project will be supported by TUScholarShare (https://scholarshare.temple.edu/), the institutional repository for Temple University. This is a repository service that is managed by the Temple University Libraries and uses Open Repository, an enhanced DSpace platform that is hosted by Atmire. TUScholarShare has been developed with the intent of helping researchers comply with grant-funding agency requirements. It enables dissemination and long-term preservation and curation (management, use, and re-use) of data.

REFERENCES:
- [Background] Russell CG, Russell A. "Food" and "non-food" self-regulation in childhood: a review and reciprocal analysis. Int J Behav Nutr Phys Act. 2020 Mar 10;17(1):33. doi: 10.1186/s12966-020-00928-5. PMID 32151265